CLINICAL TRIAL: NCT06402318
Title: A Prospective, Non-interventional, Observational Clinical Validation Study to Analytically Validate the A&M Breathalyzer PROTECT Kiosk Breath Capture System.
Brief Title: Passive Detection- SARS-CoV-2 (COVID-19) A&M Breathalyzer (PROTECT Kiosk) for Operational Medicine
Acronym: COVID-19
Status: Recruiting | Type: Observational
Sponsor: The Geneva Foundation (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Level 42 AI, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C.2024.007
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-01

CONDITIONS: COVID-19; SARS CoV 2 Virus; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome
Keywords: Breathalyzer; COVID-19 detection; Diagnostic Product; Pulmonary; PROTECT Kiosk; Passive Detection
MeSH Terms: conditions — COVID-19 | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19, Flu, or RSV positive patients: Participants screened with known COVID-19, Flu or RSV positive results obtained within 48 hours of recruitment.
  Interventions: Device: A&M Breathalyzer PROTECT Kiosk
- COVID-19, Flu or RSV negative patients: Participants screened with known COVID-19, Flu or RSV negative results obtained within 48 hours of recruitment.
  Interventions: Device: A&M Breathalyzer PROTECT Kiosk

INTERVENTIONS:
Device: A&M Breathalyzer PROTECT Kiosk — The A&M Breathalyzer PROTECT Kiosk will collect the mass spectrum breath readings from each participant, scan speed, and will autoanalyze noise and scan thresholds and sensitivity data.
  Other Names: Breathalyzer

SUMMARY:
The primary objective of this effort will be to optimize and operationalize innovative passive surveillance systems and in parallel, the effort will identify, evaluate, and transition groundbreaking new technologies in diagnostics for operationalization.

To meet the objective and execute the deliverables for this program of effort, the A&M Breathalyzer PROTECT Kiosk will be tested, modified and validated at Brooke Army Medical Center (BAMC). The collaborative efforts between the PI, Dr. Michael Morris at BAMC and Co-Investigator Dr. Tony Yuan at USU- Center for Biotechnology (4D Bio3) will assess the passive detection technology and provide a capability survey of use-case scenarios for different operational settings.

Goals:

1. Optimization and operationalize the A&M Breathalyzer PROTECT Kiosk, portable mass spectrometer (MS) Detector for Deployment in Military Operational Medicine Environments. The Breathalyzer will be deployed to BAMC to test its detection capabilities of COVID-19 among symptomatic and asymptomatic COVID-19 carrier vs. those not infected compared to gold standard RT-PCR.
2. Evaluate the passive sensing, breath capture system, built within the A&M Breathalyzer PROTECT Kiosk. The conversion of the active breath capture system, currently requires a straw that the subject breaths into, where then a series of sensors built in the Breathalyzer would automatically sample the exhaled breath within proximity for recent COVID-19 exposure. This task would conclude with a set of sensors and sensor inputs that would be analyzed by the Atomic AI platform built in the device. Field testing at BAMC is planned to determine the level of detection and discrimination for sensor combinations to SARS-CoV2 components and biomarkers detected. This testing would update the Atomic AI algorithm, within the device, to understand the accuracy of positive detection and the resulting sensitivities.

DETAILED DESCRIPTION:
Emerging acute respiratory diseases (ARDs) pose a significant threat for the US military, especially among those in training environments where crowded living conditions and demanding multi-factorial stresses exacerbate infection exposure and suppress immunity, respectively. Consequently, ARD rates are routinely reported higher in recruits than older military personnel, which have a detrimental effect on operational readiness. Although significant steps, such as surveillance and vaccine programs, have been taken to minimize the impact that ARDs have on military recruits and newly mobilized troops, hospitalizations among recruits still exceeds that of comparable civilian population in the United States by at least 3- to 4-folds, accounting for almost 30% of all infectious disease associated hospitalizations. In 2018, respiratory infections like respiratory syncytial virus (RSV), accounted for an estimated 50,000 medical encounters affecting about ~35,000 recruits that resulted in 1,000 hospital bed days leading to significant loss in training time and cost. In addition to annual respiratory infections, the on-going COVID-19 numbers rising again, continues to threaten to further degrade operational readiness. Thus, inexpensive, rapid, and more reliable diagnostics are continually required to better treat and prevent ARDs to preserve military readiness and decrease disability adjusted life years.

Current CLIA laboratory diagnostic procedures, such Enzyme Linked Immunosorbent Assay (ELISA), Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), and bacterial cultures, are costly, time-consuming, and operator sensitive. It has become apparent that during the COVID-19 pandemic, these approaches were and continue to be insufficient in meeting diagnostic needs as they are difficult to scale-up and lack logistical flexibility. Furthermore, due to the invasive nature of active clinical sampling, there is a critical need for accurate and rapid passive surveillance as to screen for SARS-CoV-19 as well as other hazardous chemical and biological agents. To address this capability gap, the current project will: 1) modify and operationalize existing innovative passive surveillance systems that can be deployed in the near-term; 2) leverage revolutionary technologies that will enhance current diagnostic systems to meet mid- and far-term gaps in CBRNE gaps.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic and symptomatic individuals 18 years and older
* Receiving standard COVID-19, Flu and/or RSV screening and testing at BAMC
* Do not have to be diagnosed with SARS-CoV-19 (COVID-19) but only be screened
* Ability to understand consent

Exclusion Criteria:

* Any individual under age of 18
* Anyone unable to comply (or be assisted) with study procedures
* Anyone not able to provide temperature thermal scan, and/or perform exhaled breath for approximately 8 seconds

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic and symptomatic individuals age 18 and older undergoing COVID-19, Flu and/or RSV screening and testing at BAMC, with and without COVID-19.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Concentration on optimization and operationalizing the A&M Breathalyzer PROTECT Kiosk | Enrollment through to study completion (min 48hrs through to 12 months)
  Optimization and operationalize the A&M Breathalyzer PROTECT Kiosk, to test its detection capabilities of COVID-19, Flu, and/or RSV among symptomatic and asymptomatic COVID-19, Flu or RSV carrier vs. those not infected compared to gold standard RT-PCR.
Concentration on evaluating the passive sensing, breath capture system built within the A&M Breathalyzer PROTECT Kiosk. | Enrollment through to study completion (min 48hrs through to 12 months)
  This evaluation would conclude with a set of sensors and sensor inputs that would be analyzed by the Atomic AI platform built in the device. Field testing at BAMC is planned to determine the level of detection and discrimination for sensor combinations to SARS-CoV2 components and biomarkers detected. This testing would update the Atomic AI algorithm, within the device, to understand the accuracy of positive detection and the resulting sensitivities.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Yuan, PhD, Principal Investigator — Uniformed Services University of the Health Sciences (USUHS); Michael Morris, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson JC. Measuring breath acetone for monitoring fat loss: Review. Obesity (Silver Spring). 2015 Dec;23(12):2327-34. doi: 10.1002/oby.21242. Epub 2015 Nov 2. PMID 26524104
- [Background] Grassin-Delyle S, Roquencourt C, Moine P, Saffroy G, Carn S, Heming N, Fleuriet J, Salvator H, Naline E, Couderc LJ, Devillier P, Thevenot EA, Annane D; Garches COVID-19 Collaborative Group RECORDS Collaborators and Exhalomics(R) Collaborators. Metabolomics of exhaled breath in critically ill COVID-19 patients: A pilot study. EBioMedicine. 2021 Jan;63:103154. doi: 10.1016/j.ebiom.2020.103154. Epub 2020 Dec 4. PMID 33279860
- [Background] Zamora-Mendoza BN, Diaz de Leon-Martinez L, Rodriguez-Aguilar M, Mizaikoff B, Flores-Ramirez R. Chemometric analysis of the global pattern of volatile organic compounds in the exhaled breath of patients with COVID-19, post-COVID and healthy subjects. Proof of concept for post-COVID assessment. Talanta. 2022 Jan 1;236:122832. doi: 10.1016/j.talanta.2021.122832. Epub 2021 Sep 2. PMID 34635222
- [Background] van Keulen KE, Jansen ME, Schrauwen RWM, Kolkman JJ, Siersema PD. Volatile organic compounds in breath can serve as a non-invasive diagnostic biomarker for the detection of advanced adenomas and colorectal cancer. Aliment Pharmacol Ther. 2020 Feb;51(3):334-346. doi: 10.1111/apt.15622. Epub 2019 Dec 20. PMID 31858615